CLINICAL TRIAL: NCT01709266
Title: A Randomized, Placebo-controlled, Double Blind Volunteer Study Into the Effect of Probiotics on Gastroenteritis Caused by an Attenuated E. Coli.
Brief Title: The Effect of Probiotics on E. Coli-induced Gastroenteritis
Acronym: PROTETEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NL40301.081.12
Record Dates: First submitted 2012-10-11; First posted 2012-10-18 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Gastroenteritis; Bacterial Infection; Diarrhea
MeSH Terms: conditions — Gastroenteritis; Bacterial Infections; Diarrhea | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Experimental): Capsule containing 5x10E9 CFU probiotics. Twice daily for 2 weeks.
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Capsule containing carrier material powder of identical appearance. Twice daily for 2 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics
  Arms: Probiotics
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Background:

The incidence of gastrointestinal infections is very high. In Western countries at least 30% of the population suffers from at least one food-borne infection per year. Mostly because of the problem of antibiotic resistance, more emphasis is put on prevention of infections. One of the possibilities is to strengthen human resistance to gut infections by consumption of probiotics. A specific blend of probiotic lactic acid bacteria (Lactobacillus helveticus Rosell-52, Lactobacillus rhamnosus Rosell-11, Bifidobacterium longum Rosell-175) and a probiotic yeast (Saccharomyces boulardii), improved stool consistency and shortened the duration of diarrhea in a rat model of E.coli-induced diarrhea. These probiotics showed synergistic effects compared with administration of solely S. boulardii or a mixture of L. helveticus Rosell-52, L. rhamnosus Rosell-11, B. longum Rosell-175. Consumption of S. boulardii and a combination of L. helveticus Rosell-52, L. rhamnosus Rosell-11 reduced diarrhea in humans.

Aim:

To study whether probiotics improves the resistance of humans to enterotoxigenic E. coli (ETEC).

Study design:

The PROTETEC study is a parallel, double-blind, placebo-controlled 4-weeks intervention with probiotics in healthy volunteers. In this study, the effect of probiotic intervention vs placebo on several infection markers in response to an ETEC challenge is investigated. Participants will be randomly assigned to the probiotic or placebo group (n=30 per group). Subjects will be instructed to maintain their usual pattern of physical activity and their habitual food intake, but to standardize their dietary calcium intake. After an adaptation period of 2 weeks, subjects will be orally infected with a live, but attenuated, ETEC vaccine (strain E1392-75-2A; collection NIZO food research; dose 10E10 CFU). Before and after infection, a diary will be kept to record all food and drinks consumption (2x2 days) to assess the habitual dietary intake, as well as for daily recording of bowel habits and frequency and severity of gastrointestinal complaints. The following biological samples will be collected: 4x10 ml venous blood, a single fecal bolus (for screening) and 7x24 hrs feces. Blood is sampled for immune response analyses and the fecal samples are collected to quantify several infection- and immune system markers, to determine probiotic excretion, and to verify dietary calcium intake.

Study population:

Healthy males of 20-55 yrs of age.

Interventions:

Probiotics (capsules containing freeze-dried powder, probiotic dose per capsule 5x10E9 CFU; twice daily) or placebo (capsules with carrier material powder of identical appearance)

Primary outcomes:

Fecal ETEC excretion and severity of diarrhea (quantified by fecal output per day).

Secondary outcomes:

Serum immune response to ETEC, self-reported stool consistency scores and gastrointestinal complaints, relative fecal wet weight.

Tertiary outcomes:

sIgA and calprotectin in feces, probiotic persistence and levels of opportunistic pathogens in the endogenous microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male
* Age 20-55 yrs
* Availability of internet connection
* Willingness to replace habitual dairy product intake with the supplied low-calcium soy products
* Willingness to abstain from products with high amounts of prebiotic fibers and from products with probiotics (except for the supplied one) starting 1 month prior to study start
* Willingness to give blood donation from 1 month before the start of the experiment and during the entire experimental period.

Exclusion Criteria:

* Current or previous underlying disease of the GI tract, liver, bile bladder, kidney, thyroid gland (self-reported)
* Allergy to milk products or lactose intolerance (self-reported), since the capsules may contain milk traces from culture media
* Allergy to soy products (self-reported)
* Use of antibiotics, norit, laxatives (up till 6 months prior to inclusion), cholestyramine, acid burn inhibitors or immune suppressive agents (up till 3 months prior to inclusion), and pre- and probiotics (up till 1 month prior to inclusion).
* High titer serum antibodies against ETEC (10 ml blood sample collected at screening)
* Vegetarians
* Vegans
* Heavy alcohol use (>4 consumptions/day or >20/week)
* Drug use

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Fecal ETEC excretion curve over time as marker of the colonization resistance | Fecal ETEC excretion measured 1-2 days before ETEC infection, and on day 1, 2, 3, 4, 7 and 15 after infection.
  The curve of fecal ETEC excretion over time is compared between verum and placebo group.
Total daily fecal output curve over time as marker of diarrhea | Daily fecal output is measured 1-2 days before ETEC infection (baseline), and on day 1, 2, 3, 4, 7 and 15 after infection.
  The curve of daily fecal output over time is compared between verum and placebo group.

SECONDARY OUTCOMES:
Bowel habits | Scored daily in a diary during 4 weeks, starting at the day of dietary intervention until 2 weeks after ETEC infection.
Frequency and severity of gastrointestinal symptoms | Scored daily by VAS scores in a diary during 4 weeks, starting at the day of dietary intervention until 2 weeks after ETEC infection.
Diarrhea severity | 1-2 days before ETEC infection, and on day 1, 2, 3, 4, 7 and 15 after infection.
  Measured by fecal dry weight excretion and % fecal dry weight.
Specific serum antibody response to CFA-II | Before and at day 3 and 15 after ETEC infection.

OTHER OUTCOMES:
Opportunistic pathogens in feces | 1-2 days before ETEC infection, and on selected time points after infection (day 1, 2, 3, 4, 7 or 15, depending on results of primary and secondary outcomes).
  Measurement of tertiary study outcomes will depend on the results of the primary and secondary study outcomes.
Calprotectin in feces | 1-2 days before ETEC infection, and on selected time points after infection (day 1, 2, 3, 4, 7 or 15, depending on results of primary and secondary outcomes).
  Measurement of tertiary study outcomes will depend on the results of the primary and secondary study outcomes.
Total faecal sIgA | 1-2 days before ETEC infection, and on seleceted time points after infection (day 1, 2, 3, 4, 7 or 15, depending on results of primary and secondary outcomes).
  Measurement of tertiary study outcomes will depend on the results of the primary and secondary study outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- NIZO Food Research, Ede, Utrecht, Netherlands

REFERENCES:
- [Result] Ten Bruggencate SJ, Girard SA, Floris-Vollenbroek EG, Bhardwaj R, Tompkins TA. The effect of a multi-strain probiotic on the resistance toward Escherichia coli challenge in a randomized, placebo-controlled, double-blind intervention study. Eur J Clin Nutr. 2015 Mar;69(3):385-91. doi: 10.1038/ejcn.2014.238. Epub 2014 Nov 5. PMID 25369827